CLINICAL TRIAL: NCT00925444
Title: Medical and Economic Evaluation of FORESEAL Versus the Current Therapeutic Approach (Stapling Alone or Associated With Tissue Sealant) in Terms of Air Leakage Duration After Lung Resection for Cancer.
Brief Title: Staple-line Reinforcement for Prevention of Pulmonary Air Leakage
Acronym: SPIRAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P080204; IDRCB 2008-A01386-49
Record Dates: First submitted 2009-06-19; First posted 2009-06-22 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2009-01

CONDITIONS: Lung Neoplasms; Pulmonary Surgical Procedures; Surgical Staplers; Tissue Adhesives; Chest Tubes
Keywords: Absorbable implants; Humans; Alginates; Pneumonectomy/methods; Pneumonectomy/instrumentation; Surgical Stapling; Thoracic surgery; Tissue Adhesives; Prospective studies
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FOREseal (Experimental)
  Interventions: Device: FOREseal
- Stapling (Active Comparator)
  Interventions: Device: Stapling

INTERVENTIONS:
Device: FOREseal — a pair of alginate sleeves for linear cutting staplers used in lung surgery
  Arms: FOREseal
Device: Stapling — Stapling alon or associated with sealants
  Arms: Stapling

SUMMARY:
The aim of this study is to compare the efficacy of FORESEAL with stapling alone or associated with tissue sealant or glue in terms of air leakage duration after lung resection for cancer.

Hypothesis: to show a significant difference of 1 day in the average duration of air leakage between the 2 groups with a standard deviation of 3 (α =0.05 and β=0.10).

DETAILED DESCRIPTION:
Air leaks continue to be the most common complication after pulmonary resection even using a stapling device. Double chest tubes after lobectomy is a well established method for drainage of the pleural cavity to allow adequate expansion of the remaining lung.

FORESEAL has been developed to reduce air leaks by buttressing the staple line. It is a absorbable vegetal biopolymer in the form of sleeves, CE marked and indicated for prevention of air leakage after pulmonary resection with stapling device. It acts as a suture reinforcement as well as a sealant thanks to its jellification.

Sealants are also commonly used in addition to stapling to prevent air leakage. The aim of this study is to compare the efficacy of FORESEAL with stapling alone or associated with sealants.

This is a multi centre, prospective controlled and randomised clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years old or over.
* Patient that undergoes a lobectomy or bilobectomy for lung cancer,
* Patient presenting an incomplete fissure, requiring stapling of at least 50% of the fissure and/or an emphysematous lung at the fissure point, requiring stapling.
* Patient that has signed the informed consent before the operation.
* Patient that benefits from a social security regime.

Exclusion Criteria:

* Patient with history of thoracotomy on the side operated on.
* Patient with severe pleural infection and/or infection of parenchyma.
* Presence of air leakage after liberation of lung in cases of pleural symphysis.
* Patient pregnant, giving birth or nursing.
* Patient presenting a contra indication to the aerostatic products used.
* Patient already participating in biomedical research.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2009-06; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Air leak (presence or absence of bubbles) will be assessed from T0: one hour after extubation, and then twice daily (morning and evening). The mean duration of post-operative air leakage will be calculated from T0 to the last day air leak observed. | from T0 to the last day air leak observed

SECONDARY OUTCOMES:
Incidence of patients presenting prolonged air leakage (lasting more than 5 days). Average duration of drainage Incidence of patients without any air leakage at 24 hours after surgery Post-operative complications Nature and costs of treatments | withing the first one year after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jean François REGNARD, PhD, Principal Investigator — Centre Hospitalier Hotel Dieu
Locations (1):
- Assistance Publique Hopitaux de Paris, Paris, France

REFERENCES:
- [Background] Fleisher AG, Evans KG, Nelems B, Finley RJ. Effect of routine fibrin glue use on the duration of air leaks after lobectomy. Ann Thorac Surg. 1990 Jan;49(1):133-4. doi: 10.1016/0003-4975(90)90371-c. PMID 2297261
- [Background] Macchiarini P, Wain J, Almy S, Dartevelle P. Experimental and clinical evaluation of a new synthetic, absorbable sealant to reduce air leaks in thoracic operations. J Thorac Cardiovasc Surg. 1999 Apr;117(4):751-8. doi: 10.1016/S0022-5223(99)70296-5. PMID 10096971
- [Background] Porte HL, Jany T, Akkad R, Conti M, Gillet PA, Guidat A, Wurtz AJ. Randomized controlled trial of a synthetic sealant for preventing alveolar air leaks after lobectomy. Ann Thorac Surg. 2001 May;71(5):1618-22. doi: 10.1016/s0003-4975(01)02468-7. PMID 11383810
- [Background] Wain JC, Kaiser LR, Johnstone DW, Yang SC, Wright CD, Friedberg JS, Feins RH, Heitmiller RF, Mathisen DJ, Selwyn MR. Trial of a novel synthetic sealant in preventing air leaks after lung resection. Ann Thorac Surg. 2001 May;71(5):1623-8; discussion 1628-9. doi: 10.1016/s0003-4975(01)02537-1. PMID 11383811
- [Background] Fabian T, Federico JA, Ponn RB. Fibrin glue in pulmonary resection: a prospective, randomized, blinded study. Ann Thorac Surg. 2003 May;75(5):1587-92. doi: 10.1016/s0003-4975(02)04994-9. PMID 12735583
- [Background] Thomas P, Massard G, Porte H, Doddoli C, Ducrocq X, Conti M. A new bioabsorbable sleeve for lung staple-line reinforcement (FOREseal): report of a three-center phase II clinical trial. Eur J Cardiothorac Surg. 2006 Jun;29(6):880-5. doi: 10.1016/j.ejcts.2006.01.067. Epub 2006 May 3. PMID 16675257
- [Background] Abolhoda A, Liu D, Brooks A, Burt M. Prolonged air leak following radical upper lobectomy: an analysis of incidence and possible risk factors. Chest. 1998 Jun;113(6):1507-10. doi: 10.1378/chest.113.6.1507. PMID 9631785
- [Background] Stephan F, Boucheseiche S, Hollande J, Flahault A, Cheffi A, Bazelly B, Bonnet F. Pulmonary complications following lung resection: a comprehensive analysis of incidence and possible risk factors. Chest. 2000 Nov;118(5):1263-70. doi: 10.1378/chest.118.5.1263. PMID 11083673
- [Background] Varela G, Jimenez MF, Novoa N, Aranda JL. Estimating hospital costs attributable to prolonged air leak in pulmonary lobectomy. Eur J Cardiothorac Surg. 2005 Feb;27(2):329-33. doi: 10.1016/j.ejcts.2004.11.005. PMID 15691691
- [Background] Mouritzen C, Dromer M, Keinecke HO. The effect of fibrin glueing to seal bronchial and alveolar leakages after pulmonary resections and decortications. Eur J Cardiothorac Surg. 1993;7(2):75-80. doi: 10.1016/1010-7940(93)90184-d. PMID 8442983
- [Background] Wong K, Goldstraw P. Effect of fibrin glue in the reduction of postthoracotomy alveolar air leak. Ann Thorac Surg. 1997 Oct;64(4):979-81. doi: 10.1016/s0003-4975(97)00820-5. PMID 9354513
- [Background] Tansley P, Al-Mulhim F, Lim E, Ladas G, Goldstraw P. A prospective, randomized, controlled trial of the effectiveness of BioGlue in treating alveolar air leaks. J Thorac Cardiovasc Surg. 2006 Jul;132(1):105-12. doi: 10.1016/j.jtcvs.2006.02.022. PMID 16798309
- [Background] Rami R, Mateu M. Surgical sealant for preventing air leaks after pulmonary resections in patients with lung cancer. Cochrane Database Syst Rev. 2001;(4):CD003051. doi: 10.1002/14651858.CD003051. PMID 11687173
- [Background] Belboul A, Dernevik L, Aljassim O, Skrbic B, Radberg G, Roberts D. The effect of autologous fibrin sealant (Vivostat) on morbidity after pulmonary lobectomy: a prospective randomised, blinded study. Eur J Cardiothorac Surg. 2004 Dec;26(6):1187-91. doi: 10.1016/j.ejcts.2004.08.009. PMID 15541982